CLINICAL TRIAL: NCT00648076
Title: Single-Dose Food In Vivo Bioequivalence Study of Divalproex Sodium Extended-Release Tablets (500 mg; Mylan) to Depakote ER® Tablets (500 mg; Abbott) in Healthy, Adult Male Volunteers
Brief Title: Food Study of Divalproex Sodium Extended-Release Tablets 500 mg to Depakote ER® Tablets 500 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DIVA-0381
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
MeSH Terms: interventions — Valproic Acid

ARMS (2):
- 1 (Experimental): Divalproex Sodium Extended-Release Tablets 500 mg
  Interventions: Drug: Divalproex Sodium Extended-Release Tablets 500 mg
- 2 (Active Comparator): Depakote ER® Tablets 500 mg
  Interventions: Drug: Depakote ER® Tablets 500 mg

INTERVENTIONS:
Drug: Divalproex Sodium Extended-Release Tablets 500 mg — 500mg, single dose fed
  Arms: 1
Drug: Depakote ER® Tablets 500 mg — 500mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's divalproex sodium 500 mg extended-release tablets to Abbott's Depakote ER® 500 mg tablets following a single, oral 500 mg (1 x 500 mg) dose administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male.
3. Weight: At least 60 kg (132 lbs) and within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, including vital signs, laboratory evaluation, 12-lead ECG, hepatitis B and hepatitis C tests, HIV test, and urine drug screen including amphetamine, barbiturates, benzodiazepine, cannabinoid, cocaine, opiates, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.
5. During the course of the study, from study screen until study exit, all males must use a spermicide-containing barrier method of contraception in addition to their current contraceptive device (if any). This requirement should be documented in the informed consent form.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to valproic acid or any other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Freeland, D.O., Principal Investigator — Cedra Clinical Research, LLC.
Locations (1):
- Cedra Clinical Research, LLC., Austin, Texas, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html